CLINICAL TRIAL: NCT02415075
Title: Experten-Prävention Bei gefährdeter Erwerbsfähigkeit Durch Telefonische, Motivierende Interviews Zur Unterstützung Des Selbstmanagements
Brief Title: Prevention of Reduced Employability With an Expert System With Telephone, Motivational Interviews Supporting Self-management
Acronym: EXPERTIS
Status: Completed | Type: Observational
Sponsor: Jacobs University Bremen gGmbH (Other)
Responsible Party: Principal Investigator, Prof. Dr. Sonia Lippke, Professor of Health Psychology, Jacobs University Bremen gGmbH
Other Study IDs: 060.007.15.00-3.005-JUB
Record Dates: First submitted 2015-04-02; First posted 2015-04-14 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Employability
Keywords: Return to work, state of subjective health, medical rehabilitation, motivational interviewing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: medical rehabilitation — Participants who will take part in the study are asked to fill out a questionnaire when arriving at the rehabilitation clinic and will be invited to participate in two motivational telephone interviews after six and 12 months.

SUMMARY:
The purpose of the study is to determine which factors on a personal, social and contextual level will help rehabilitation patients on returning to or continuing to work as well as to stay employable.

DETAILED DESCRIPTION:
For most people work is an integral part of their life which not only secures their life standards, but also forms the basis for social participation and personal growth. If someone's workability is limited as a result of health problems, medical rehabilitation can often help to regain strength and capabilities, and to continue to work in a productive way and remain healthy. In cooperation with the Deutsche Rentenversicherung Oldenburg-Bremen health psychologists at Jacobs University Bremen are investigating what contributes to the success of such medical rehabilitation treatments.

The focus is to understand which measures are helping people during and subsequently to their treatment in the clinic.Therefore voluntary participants will be asked to fill out a questionnaire when arriving at the rehabilitation facility and will subsequently invited to participate in two motivational telephone interviews after six and 12 months. Personal, social and contextual factors, measures and offers, as well as goals, plans and behaviors, will be taken into consideration to evaluate the effectiveness of medical rehabilitation on returning to or continuing to work.

ELIGIBILITY:
Inclusion Criteria:

* insurants of the Deutsche Rentenversicherung Oldenburg-Bremen
* with a granted medical rehabilitation stay
* sufficient knowledge of the German, Turkish or Russian language
* telephone or mobile phone connections

Exclusion Criteria:

* insurants of the Deutsche Rentenversicherung Oldenburg-Bremen who did not receive a granted stay at one of the medical rehabilitation clinics of the Deutsche Rentenversicherung Oldenburg-Bremen
* no proficient language skills (German, Turkish, Russian)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the study insurants of the Deutsche Rentenversicherung Oldenburg-Bremen with a granted medical rehabilitation treatment will be asked to fill out a questionnaire when arriving at the rehabilitation clinic as well as to take part in two subsequent telephone interviews after 6 and 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 1045 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
quality of life and life satisfaction | when arriving at the rehabilitation clinic (t1)
  self-report questionnaire (expected number of participants for the measures: 926)
change in quality of life and life satisfaction at 6 and 12 months | after the rehabilitation treatment at 6 (t2) and 12 (t3) months
  self-report (as described above two subsequent telephone interviews after 6 and 12 months)
motivation for returning to work | when arriving at the rehabilitation clinic (t1)
  self-report questionnaire
change in motivation for returning to work at 6 and 12 months | after the rehabilitation treatment at 6 (t2) and 12 (t3) months
  self-report
actual return to work | after the rehabilitation treatment at 6 (t2) months
  self-report
actual return to work | after the rehabilitation treatment at 12 (t3) months
  self-report

SECONDARY OUTCOMES:
personal goals and plans | when arriving at the rehabilitation clinic (t1)
  self-report questionnaire
change in personal goals and plans at 6 months | after the rehabilitation treatment at 6 months (t2)
  self-report
change in personal goals and plans at 12 months | after the rehabilitation treatment at 12 months (t3)
  self-report
social-cognitive variables (e.g. self-efficacy, social support) | when arriving at the rehabilitation clinic (t1)
  self-report questionnaire
social-cognitive variables (e.g. self-efficacy, social support) | after the rehabilitation treatment at 6 months (t2)
  self-report
social-cognitive variables (e.g. self-efficacy, social support) | after the rehabilitation treatment at 12 months (t3)
  self-report
physical activity level (based on IPAQ) | when arriving at the rehabilitation clinic (t1)
  self-report questionnaire
physical activity level (based on IPAQ) | after the rehabilitation treatment at 6 months (t2)
  self-report
physical activity level (based on IPAQ) | after the rehabilitation treatment at 12 months (t3)
  self-report
socio-economic and socio-demographic variables | when arriving at the rehabilitation clinic (t1)
  self-report questionnaire
socio-economic and socio-demographic variables | after the rehabilitation treatment at 6 months (t2)
  self-report
socio-economic and socio-demographic variables | after the rehabilitation treatment at 12 months (t3)
  self-report
subjective health and self-reported diagnoses | when arriving at the rehabilitation clinic (t1)
  self-report questionnaire
subjective health and self-reported diagnoses | after the rehabilitation treatment at 6 months (t2)
  self-report
subjective health and self-reported diagnoses | after the rehabilitation treatment at 12 months (t3)
  self-report
employment history | when arriving at the rehabilitation clinic (t1)
  self-report questionnaire
Questions on the expectations of the medical rehabilitation | when arriving at the rehabilitation clinic (t1)
  self-report questionnaire
Questions on the satisfaction with the medical rehabilitation treatments | after the rehabilitation treatment at 6 months (t2)
  self-report

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Lippke, Prof. Dr., Principal Investigator — Jacobs University Bremen gGmbH
Locations (1):
- Jacobs University Bremen gGmbH, Bremen, Germany

REFERENCES:
- [Derived] Rinn R, Whittal A, Kremeti E, Lippke S. The social class of orthopedic rehabilitation patients: Are there differences in subjective health, return to work motivation, and participation in aftercare interventions? Soc Sci Med. 2024 Sep;356:117152. doi: 10.1016/j.socscimed.2024.117152. Epub 2024 Jul 17. PMID 39047522